CLINICAL TRIAL: NCT00394771
Title: A Prospective, Multicenter, Double-Blinded, Randomized Study to Evaluate Bleeding Patterns in Women Using One of Three Different Doses of DR-1031 Oral Contraceptive Compared to Seasonale Oral Contraceptive Regimen
Brief Title: A Study to Evaluate Bleeding Patterns With Three Different Doses of DR-1031 Compared to Seasonale
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DR-ASC-201
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Breakthrough Bleeding
Keywords: oral contraceptives; breakthrough bleeding; spotting
MeSH Terms: conditions — Metrorrhagia | interventions — Ethinyl Estradiol-Norgestrel Combination; Seasonale

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Dose DR-1031 (Experimental): 42 days combination active tablets (20 mcg EE /150 mcg LNG) followed by 21 days combination active tablets (25 mcg EE/150 mcg LNG) followed by 21 days combination active tablets (30 mcg EE/ 150 mcg LNG) followed by 7 days of 10 mcg EE tablets.
  Interventions: Drug: DR-1031; Drug: Portia®
- Midrange Dose DR-1031 (Experimental): 21 days combination active tablets (20 mcg EE /150 mcg LNG) followed by 42 days combination active tablets (25 mcg EE/ 150 mcg LNG) followed by 21 days combination active tablets (30 mcg EE/ 150 mcg LNG) followed by 7 days of 10 mcg EE tablets.
  Interventions: Drug: DR-1031; Drug: Portia®
- High Dose DR-1031 (Experimental): 21 days combination active tablets (20 mcg EE /150 mcg LNG) followed by 21 days combination active tablets (25 mcg EE/150 mcg LNG) followed by 42 days combination active tablets (30 mcg EE/ 150 mcg LNG) followed by 7 days of 10 mcg EE tablets.
  Interventions: Drug: DR-1031; Drug: Portia®
- Seasonale (Active Comparator): 84 days of combination active tablets, each containing 30 mcg EE and 150 mcg LNG, followed by 7 days of placebo tablets.
  Interventions: Drug: Seasonale®; Drug: Portia®

INTERVENTIONS:
Drug: DR-1031 — Active therapy cycle of 84 days taking combination tablets containing ascending doses of ethinyl estradiol (EE) and 150 mcg levonorgestrel (LNG), followed by a 7-day withdrawal cycle of 10 mcg EE. The total extended cycle was 91 days and participants were to complete two extended cycles. Active therapy dosage of EE varied by treatment arm.
  Other Names: levonorgestrel/ethinyl estradiol; Quartette®
  Arms: High Dose DR-1031; Low Dose DR-1031; Midrange Dose DR-1031
Drug: Seasonale® — 84 days of combination active tablets, each containing 30 mcg EE and 150 mcg LNG, followed by 7 days of placebo tablets for two consecutive 91-day cycles.
  Other Names: levonorgestrel/ethinyl estradiol
  Arms: Seasonale
Drug: Portia® — Portia® 28 consists of 21 pink active tablets, each containing 0.15 mg of levonorgestrel and 0.03 mg of ethinyl estradiol, and seven white inert tablets. Portia was taken as a pre-study run-in medication.
  Other Names: levonorgestrel/ethinyl estradiol

SUMMARY:
This is a 4-arm study to evaluate and compare bleeding patterns between three different doses of DR-1031 oral contraceptive with Seasonale oral contraceptive. Study participants will receive physical and gynecological exams, including Pap smear. During the study, all participants will be required to complete a diary

DETAILED DESCRIPTION:
This Phase 2, prospective, multicenter, double-blinded, randomized study is designed to evaluate and compare bleeding patterns in women using one of three different doses of DR-1031 oral contraceptive with Seasonale oral contraceptive.

Patients who meet all study entrance criteria will be randomly assigned to one of four treatment groups,

The overall study duration will be approximately 9 months; this will include a screening period of approximately 4 weeks, a run-in period of 4 weeks, a treatment period of approximately 6 months (two,91-day cycles) and a final study visit occurring 14-21 days after completion of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Not pregnant or breastfeeding
* Agree to use back-up non-hormonal contraception for study period

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Pregnancy within the last 3 months
* Smoking >10 cigarettes per day

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 567 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Medical Monitor, Principal Investigator — Duramed Research
Locations (48):
- United States (48):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Little Rock, Arkansas
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, San Francisco, California
  - Duramed Investigational Site, Santa Ana, California
  - Duramed Investigational Site, Vista, California
  - Duramed Investigational Site, Pueblo, Colorado
  - Duramed Investigational Site, Stratford, Connecticut
  - Duramed Investigational Site, DeLand, Florida
  - Duramed Investigational Site, Jacksonville, Florida
  - Duramed Investigational Site, Melbourne, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, West Palm Beach, Florida
  - Duramed Investigational Site, Alpharetta, Georgia
  - Duramed Investigational Site, Douglasville, Georgia
  - Duramed Investigational Site, Savannah, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Meridian, Idaho
  - Duramed Investigational Site, Fort Wayne, Indiana
  - Duramed Investigational Site, Wichita, Kansas
  - Duramed Investigational Site, Baton Rouge, Louisiana
  - Duramed Investigational Site, Metairie, Louisiana
  - Duramed Investigational Site, Shreveport, Louisiana
  - Duramed Investigational Site, Riverdale, Maryland
  - Duramed Investigational Site, Kansas City, Missouri
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, North Las Vegas, Nevada
  - Duramed Investigational Site, Lebanon, New Hampshire
  - Duramed Investigational Site, Cary, North Carolina
  - Duramed Investigational Site, New Bern, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Mayfield Heights, Ohio
  - Duramed Investigational Site, Eugene, Oregon
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Charleston, South Carolina
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Hilton Head Island, South Carolina
  - Duramed Investigational Site, Jackson, Tennessee
  - Duramed Investigational Site, Austin, Texas
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Williston, Vermont

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 988 subjects were screened for participation in this study, and 567 took at least one dose of investigational product (Safety population).
Period: Overall Study
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Started | 140 (Safety population of treated participants) | 136 (Safety population of treated participants) | 143 (Safety population of treated participants) | 148 (Safety population of treated participants)
Intent to Treat (ITT) Population | 110 (At least one completed 91 day cycle of treatment) | 110 (At least one completed 91 day cycle of treatment) | 108 (At least one completed 91 day cycle of treatment) | 120 (At least one completed 91 day cycle of treatment)
Completed | 99 | 102 | 96 | 109
Not Completed | 41 | 34 | 47 | 39
Not completed — Did not meet protocol requirements | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 4 | 9 | 7
Not completed — Withdrawal by Subject | 10 | 6 | 8 | 12
Not completed — Adverse Event | 10 | 5 | 12 | 8
Not completed — Participant pregnant | 0 | 1 | 2 | 2
Not completed — Lost to Follow-up | 15 | 15 | 13 | 10
Not completed — Other | 3 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale | Total
Number analyzed (Participants) | 110 | 110 | 108 | 120 | 448
Age Continuous [Mean (Standard Deviation); unit: years] | 30.1 (6.88) | 30.5 (7.02) | 30.7 (7.61) | 30.6 (6.90) | 30.5 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 110 | 108 | 120 | 448
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 21 | 20 | 18 | 17 | 76
  Asian | 1 | 4 | 1 | 3 | 9
  Caucasian | 72 | 68 | 69 | 82 | 291
  Hispanic | 13 | 17 | 19 | 16 | 65
  Other | 3 | 1 | 1 | 2 | 7
Weight [Mean (Standard Deviation); unit: lbs] | 156.6 (28.84) | 153.6 (27.18) | 156.0 (30.79) | 151.9 (30.03) | 154.4 (29.22)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (4.13) | 25.7 (4.24) | 26.0 (4.59) | 25.5 (4.41) | 25.9 (4.35)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 114.2 (10.74) | 114.4 (10.34) | 115.6 (9.31) | 112.8 (10.23) | 114.2 (10.19)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72.3 (8.85) | 72.9 (7.46) | 71.8 (7.72) | 71.4 (8.44) | 72.1 (8.14)
Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 73.9 (9.85) | 73.7 (8.90) | 73.7 (9.17) | 71.9 (9.07) | 73.3 (9.26)
Smoking Status [Number; unit: participants]
  Current Smoker | 13 | 16 | 11 | 11 | 51
  Past Smoker | 20 | 11 | 12 | 21 | 64
  Non-Smoker | 77 | 83 | 85 | 88 | 333
Oral Contraceptive Use History [Number; unit: participants]
  Missing | 1 | 0 | 0 | 0 | 1
  Continuous User | 44 | 46 | 42 | 49 | 181
  Prior User | 44 | 45 | 49 | 52 | 190
  Fresh-Start | 21 | 19 | 17 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: Days With Bleeding and/or Spotting During Active Cycle 1 (Day 1-84)
Description: Bleeding is defined as a flow heavy enough to require sanitary protection. Spotting does not require sanitary protection.
Time Frame: Day 1-84
Population: Intent to treat (ITT) population of participants who completed the relevant pages in the patient diary.
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 110 | 110 | 108 | 120
days | 13 [0 to 67] | 13.5 [0 to 65] | 15 [0 to 69] | 15 [0 to 56]

2. Secondary Outcome: Days With Bleeding During Active Cycle 1 (Day 1-84)
Description: Bleeding is defined as a flow heavy enough to require sanitary protection.
Time Frame: Day 1-84
Population: Intent to treat (ITT) population of participants who completed the relevant pages in the patient diary.
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 110 | 110 | 108 | 120
days | 3.5 [0 to 24] | 2.5 [0 to 49] | 4 [0 to 47] | 2 [0 to 24]

3. Secondary Outcome: Days With Bleeding During Active Cycle 2 (Day 92-176)
Description: Bleeding is defined as a flow heavy enough to require sanitary protection.
Time Frame: Day 92-176
Population: Intent to treat (ITT) population of participants who were still active in the study and who completed the relevant pages in the patient diary.
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 109 | 108 | 107 | 120
days | 1 [0 to 24] | 2 [0 to 49] | 1 [0 to 27] | 2 [0 to 23]

4. Secondary Outcome: Time to First Bleeding Day
Description: Time to first bleeding day was defined as the time between the start of intervention until the first day when bleeding was heavy enough to require the use of sanitary protection.
  Data are not summarized due to limitations in the diary data and an inability to accurately determine a participant's first day of bleeding.
Time Frame: Day 1-84
Population: ITT population. However this data was not summarized due to limitations in the diary data.
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Bleeding Severity During Active Cycle 1 (Day 1-84)
Description: Bleeding is defined as a flow heavy enough to require sanitary protection. Participants recorded in the diary days when they had bleeding, and whether they considered the bleeding to be light, moderate or heavy.
  Data was not summarized due to limitations in the diary data, and an inability to accurately determine the maximum bleeding severity.
  See pre-specified analyses for Number of Moderate to Heavy Bleeding Days.
Time Frame: Day 1-84
Population: ITT population. However data was not summarized due to limitations in the diary data.
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Days With Bleeding and/or Spotting During Active Cycle 2 (Day 92-176)
Description: as for outcome 1
Time Frame: Day 92-176
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 109 | 108 | 107 | 120
days | 6 [0 to 74] | 7 [0 to 70] | 5 [0 to 74] | 6 [0 to 55]

7. Secondary Outcome: Participants With Bleeding and/or Spotting Days During the 7-day Withdrawal During Cycle 1 (Day 85-91)
Description: Participants are categorized by the duration of bleeding that occurred during the scheduled 7-day withdrawal period for Cycle 1.
Time Frame: Day 85-91
Population: Intent to treat (ITT) population of participants who completed the relevant pages in the patient diary.
Measure: Number; unit: participants
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 109 | 108 | 106 | 120
participants
  0 day | 14 | 28 | 25 | 27
  1-3 days | 36 | 17 | 27 | 18
  4-7 days | 59 | 63 | 54 | 75

8. Secondary Outcome: Participants With Bleeding and/or Spotting Days During the 7-day Withdrawal During Cycle 2 (Day 177-183)
Description: Participants are categorized by the duration of bleeding that occurred during the scheduled 7-day withdrawal period for Cycle 2.
Time Frame: Day 177-183
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 97 | 96 | 94 | 105
participants
  0 day | 15 | 20 | 23 | 21
  1-3 days | 32 | 32 | 26 | 24
  4-7 days | 50 | 44 | 45 | 60

9. Secondary Outcome: Participants Reporting Hormone-Related Symptoms During Active Cycle 1 (Day 1-84)
Description: Hormone-related symptoms include breast tenderness/pain, headache, bloating, pelvic pain, anxiety, depression, and irritability.
Time Frame: Day 1-84
Population: Intent to treat (ITT) population of participants who completed the relevant pages in the patient diary.
Measure: Number; unit: participants
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 110 | 110 | 108 | 120
participants
  Breast tenderness/pain | 58 | 57 | 50 | 64
  Headache | 83 | 84 | 86 | 92
  Bloating | 80 | 76 | 72 | 84
  Pelvic pain | 72 | 65 | 61 | 67
  Anxiety | 42 | 43 | 34 | 59
  Depression | 51 | 40 | 36 | 52
  Irritability | 72 | 69 | 66 | 78

10. Secondary Outcome: Participants Reporting Hormone-Related Symptoms During Active Cycle 2 (Day 92-176)
Description: as for outcome 9
Time Frame: Day 92-176
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 109 | 108 | 107 | 120
participants
  Breast tenderness/pain | 46 | 47 | 44 | 44
  Headache | 74 | 72 | 72 | 78
  Bloating | 64 | 64 | 57 | 70
  Pelvic pain | 58 | 57 | 45 | 57
  Anxiety | 40 | 40 | 31 | 47
  Depression | 41 | 39 | 30 | 44
  Irritability | 55 | 63 | 54 | 65

11. Secondary Outcome: Participants Reporting Hormone-Related Symptoms During the 7-day Withdrawal Cycle 1 (Day 85-91)
Description: as for outcome 9
Time Frame: Day 85-91
Population: Intent to treat (ITT) population of participants who completed the relevant pages in the patient diary.
Measure: Number; unit: participants
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 110 | 110 | 108 | 120
participants
  Breast tenderness/pain | 33 | 28 | 17 | 33
  Headache | 57 | 50 | 57 | 50
  Bloating | 61 | 51 | 46 | 62
  Pelvic pain | 50 | 49 | 37 | 53
  Anxiety | 26 | 17 | 14 | 22
  Depression | 25 | 21 | 17 | 23
  Irritability | 44 | 43 | 23 | 36

12. Secondary Outcome: Participants Reporting Hormone-Related Symptoms During the 7-day Withdrawal Cycle 2 (Day 177-183)
Description: as for outcome 9
Time Frame: Day 177-183
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 97 | 96 | 94 | 105
participants
  Breast tenderness/pain | 29 | 25 | 15 | 25
  Headache | 39 | 42 | 37 | 48
  Bloating | 51 | 53 | 38 | 60
  Pelvic pain | 52 | 42 | 31 | 51
  Anxiety | 21 | 22 | 13 | 22
  Depression | 18 | 21 | 15 | 17
  Irritability | 39 | 37 | 25 | 39

13. Other Pre Specified Outcome: Number of Moderate to Heavy Bleeding Days During Active Cycle 1 (Day 1-84)
Description: Bleeding is defined as a flow heavy enough to require sanitary protection. Participants recorded in the diary days when they had bleeding, and whether they considered the bleeding to be light, moderate or heavy.
Time Frame: Day 1-84
Population: Intent to treat (ITT) population of participants who completed the relevant pages in the patient diary.
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 110 | 110 | 108 | 120
days | 0 [0 to 12] | 0 [0 to 19] | 0 [0 to 16] | 0 [0 to 21]

14. Other Pre Specified Outcome: Number of Moderate to Heavy Bleeding Days During Active Cycle 2 (Day 92-176)
Description: as for outcome 13
Time Frame: Day 92-176
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Number analyzed (Participants) | 109 | 108 | 107 | 120
days | 0 [0 to 11] | 0 [0 to 13] | 0 [0 to 8] | 0 [0 to 7]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 256 (longest treatment plus 14 days)
Arm/Group | Low Dose DR-1031 | Midrange Dose DR-1031 | High Dose DR-1031 | Seasonale
Serious Adverse Events (participants affected / at risk) | 1/140 | 2/136 | 3/143 | 5/148
Other Adverse Events (participants affected / at risk) | 61/140 | 44/136 | 49/143 | 53/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose DR-1031 (N=140) | Midrange Dose DR-1031 (N=136) | High Dose DR-1031 (N=143) | Seasonale (N=148)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Polytraumatism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose DR-1031 (N=140) | Midrange Dose DR-1031 (N=136) | High Dose DR-1031 (N=143) | Seasonale (N=148)
Headache (Nervous system disorders) | 19 | 19 | 23 | 19
Migraine (Nervous system disorders) | 2 | 7 | 1 | 2
Nasopharyngitis (Infections and infestations) | 15 | 7 | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 5 | 9
Sinusitis (Infections and infestations) | 10 | 6 | 2 | 6
Urinary tract infection (Infections and infestations) | 8 | 1 | 5 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 13 | 6 | 5 | 7
Weight increased (Investigations) | 6 | 4 | 9 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized or published in any form to cooperative publication without prior, written consent of sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.